CLINICAL TRIAL: NCT06066190
Title: The Effect of Web-Based Education Given to Midwives and Nurses on Their Knowledge Levels Regarding ERAS Protocols Applied in Gynecological and Obstetric Surgery
Brief Title: Web-Based Education on ERAS Protocols Applied in Gynecological and Obstetric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aslı SİS ÇELİK, Associate Professor, Ataturk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: aslı15
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: ERAS
MeSH Terms: interventions — Obstetric Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: web based training (Experimental): Web-Based Training will be given to midwives and nurses on ERAS Protocols Applied in Gynecological and Obstetric Surgery. The training will last 6 weeks and they will be asked to watch a training video every week.
  Interventions: Other: Web-Based Training on ERAS Protocols Applied in Gynecological and Obstetric Surgery

INTERVENTIONS:
Other: Web-Based Training on ERAS Protocols Applied in Gynecological and Obstetric Surgery — Web-Based Training will be given to Midwives and Nurses on ERAS Protocols Applied in Gynecological and Obstetric Surgery. The training will last 6 weeks and they will be asked to watch a training video every week.

SUMMARY:
In this research, a pretest-posttest single group quasi-experimental model will be used. The study will be conducted to determine the effect of web-based training given to midwives and nurses on their level of knowledge regarding ERAS protocols applied in gynecological and obstetric surgery. It will be carried out with midwives and nurses working in the Gynecology and Obstetrics units (clinic, operating room, delivery room) of a state hospital located in a city in the east of Turkey. As an initiative, "web-based training on ERAS protocols applied in gynecological and obstetric surgery" will be provided to Midwives and Nurses. The pre-test data of the research will be collected face to face by the researcher between 1-30 November 2023 with midwives and nurses working in the relevant units in the relevant hospital, information will be given about the research and midwives and nurses who meet the sampling criteria will be given a "Descriptive Characteristic Form" and "ERAS Knowledge Test". will be implemented. Educational program; It will be implemented over a period of 1.5 months through a website specially prepared for midwives and nurses. After the training is completed, the "ERAS Protocols Applied in Gynecological and Obstetric Surgery" booklet will be given. In the web-based training system, the training will be uploaded 6 times with an interval of 1 week for midwives and nurses to listen to, and after the training is completed (January 15-21, 2024), the "Descriptive Feature Form" and "ERAS Knowledge Test" will be re-applied and post-test data will be collected.

DETAILED DESCRIPTION:
In this research, a pretest-posttest single group quasi-experimental model will be used. The study will be conducted to determine the effect of web-based training given to midwives and nurses on their level of knowledge regarding ERAS protocols applied in gynecological and obstetric surgery. It will be carried out with midwives and nurses working in the Gynecology and Obstetrics units (clinic, operating room, delivery room) of a state hospital located in a city in the east of Turkey.

The population of the research will consist of 88 midwives and nurses working in the gynecology and obstetrics units of the relevant hospital (clinic, operating room, delivery room). A pre-study power analysis was conducted using the "G Power-3.1.9.2 Program" according to the paired t test, which will be used to compare the pre-test and post-test knowledge levels of the midwives and nurses to be included in the study. It was determined that a total of 45 midwives and nurses should be included in the study with a medium effect size (0.5), 5% margin of error and 95% confidence interval.

The sample of the research will include 55 midwives and nurses (10 additional person will be taken considering the possibility of data loss), who are selected from the population by improbable random sampling method, meet the research criteria and agree to participate in the research. As an initiative, "web-based training on ERAS protocols applied in gynecological and obstetric surgery" will be provided to Midwives and Nurses.

The pre-test data of the research will be collected face to face by the researcher between 1-30 November 2023 with midwives and nurses working in the relevant units in the relevant hospital, information will be given about the research and midwives and nurses who meet the sampling criteria will be given a "Descriptive Characteristic Form" and "ERAS Knowledge Test". will be implemented. Educational program; It will be implemented over a period of 1.5 months through a website specially prepared for midwives and nurses. After the training is completed, the "ERAS Protocols Applied in Gynecological and Obstetric Surgery" booklet will be given. In the web-based training system, the training will be uploaded 6 times with an interval of 1 week for midwives and nurses to listen to, and after the training is completed (January 15-21, 2024), the "Descriptive Feature Form" and "ERAS Knowledge Test" will be re-applied and post-test data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Working in gynecology and obstetrics-related units
* Not receiving information about ERAS protocols from any source before.
* Volunteering to participate in the study

Exclusion Criteria:

* Leaving the study at any stage of the study
* Not watching the training videos that participants were required to watch in the study.
* Not filling out the online survey for post-test data at the end of the training.
* Obtain information about the ERAS Protocol from somewhere other than the Web-based training to be given within the scope of the research.

Max Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-01-21 (Estimated)

PRIMARY OUTCOMES:
Knowledge levels of Midwives and Nurses regarding ERAS Protocols Applied in Gynecological and Obstetric Surgery | 1 month
  Pre-test knowledge levels of Midwives and Nurses regarding ERAS Protocols Applied in Gynecological and Obstetric Surgery, will obtain before the intervention by applying the ERAS knowledge test. 1 point will be received for a correct answer and 0 points will be received for an incorrect answer to each question. High scores will indicate that midwives and nurses have a high level of knowledge about ERAS Protocols Applied in Gynecological and Obstetric Surgery.

SECONDARY OUTCOMES:
Change in Midwives' and Nurses' Knowledge Levels About ERAS Protocols Applied in Gynecological and Obstetric Surgery | 2 months
  The difference between the ERAS knowledge test and pre-test and post-test score averages of midwives and nurses receiving web-based training will be obtained. In the ERAS knowledge test, 1 point will be given for a correct answer to each question and 0 point will be given for an incorrect answer. High scores will indicate that midwives and nurses have a high level of knowledge about ERAS Protocols Applied in Gynecological and Obstetric Surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Aslı SİS ÇELİK, Study Director — Ataturk University